CLINICAL TRIAL: NCT00507286
Title: Efficacy and Safety Study of Using Oral Sildenafil and Intracavernosal Alprostadil Injection as a Combined Pharmacotherapy for Men With Difficult to Treat Erectile Dysfunction.
Brief Title: Efficacy and Safety Study of Combined Oral and Injection Therapy for Erectile Dysfunction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Keogh Institute for Medical Research (Other)
Responsible Party: Professor Bronwyn Stuckey, Keogh Institute for Medical Research
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Protocol No. 2005-166; Australia CTN: 2007/288
Record Dates: First submitted 2007-07-25; First posted 2007-07-26 (Estimated); Last update posted 2009-01-28 (Estimated); Status verified 2007-07

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction | interventions — Alprostadil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: combination of various doses of sildenefil and alprostadil

SUMMARY:
Erectile dysfunction (ED or impotence) is a common medical condition affecting many men world wide. The most commonly used treatment for ED are oral medications like Viagra (sildenafil), Levitra (vardenafil) and Cialis (tadalafil). If these are not effective the use of an injection into the penis (intracavernosal injection or ICI) is necessary. However in some men neither of these therapies is successful.

Hypothesis: An adequate erection may be achieved in men with difficult-to-treat erectile dysfunction, when they are treated with a therapy of combination of tablet and penile injection, when a single treatment therapy has failed for these men.

Aim of the study is to test the safety and efficacy of a combination of Viagra and Caverjet Impulse in a group of men who had failed to achieve an adequate response to the maximum recommended dose of either Viagra, Cialis or Levitra and Caverjet Impulse, when these treatments were used alone.

20 men with difficult to treat ED will be given oral medication, intracavernosal therapy or the combination in a single-blind randomised study.

Informed consent will be signed prior to any study procedures being carried out. All participants are 'blinded' to their study treatments. Participants who have satisfactory response to any of the tablets or penile injections, will be excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 20 years and over
* History of ED for at least 6 months
* IIEF score <26
* Failure to achieve an adequate response to the maximum recommended therapeutic dose of an approved ED treatments, when either of these treatments was used alone.

Exclusion Criteria:

* Concurrent treatment with nitrate-containing medications
* Significant cardiac, hepatic, renal or respiratory dysfunction
* Systolic blood pressure of less than 100mm Hg
* Myocardial infarction, serious cardiac arrhythmia, cardiac surgery, or stroke within the last 6 months
* Significant penile fibrosis, curvature or infection
* Reported significant side effects of using PDE5 inhibitors or alprostadil
* Hypersensitivity to PDE5 inhibitors or alprostadil

Min Age: 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2007-05; Primary Completion 2008-09 (Estimated); Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Sexual Encounter Profile SEP2 and SEP3

CONTACTS AND LOCATIONS:
Overall Officials: Bronwyn G STUCKEY, MBBS,FRACP, Principal Investigator — Keogh Institute for Medical Research
Locations (1):
- Keogh Institute for Medical Research, 'A' Block 3rd Floor, QE II Medical Centre, Nedlands, Perth, Western Australia, Australia